CLINICAL TRIAL: NCT00142077
Title: Health Promotion in the Workplace Using Personally Controlled Health Records
Brief Title: Electronic Health Records for Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1 R01 CDC 000065-01
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2006-01

CONDITIONS: Influenza
Keywords: Influenza; Electronic health record; Behavior modification
MeSH Terms: conditions — Influenza, Human | interventions — Electronic Health Records

INTERVENTIONS:
Device: Electronic health record and messaging system

SUMMARY:
The purpose of this study is to determine whether personally controlled electronic health records can be used for health promotion in a workplace setting.

DETAILED DESCRIPTION:
In response to the call for research of the new Health Protection Research Initiative at the Centers for Disease Control and Prevention (CDC), we propose to adapt newly mature informatics technology to shift the paradigm for health alerting and health promotion in the workplace. The goal is to firmly ground these activities on real time information collected from and delivered to employees, in an interactive, secure, electronic environment. We will study influenza prevention and control, an archetype of public health practice requiring surveillance, communication, and timely influence of health-related behaviors. Complex information gleaned from surveillance will be processed, translated and provided to employees. The goal is to provide employees with timely, individualized health promotion messages to improve their knowledge, attitudes and beliefs regarding influenza and to increase the rate of seasonal influenza immunization for them and their household members. The approach will be evaluated in a group randomized design at several worksites of a major corporation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a part-time or full-time employee at a major corporation.
2. The subject is eighteen years of age or older.
3. The subject is comfortable reading and writing in English.
4. The subject has reliable internet access at home, at school, or at work.
5. The subject uses email regularly (i.e. at least once every 2 days)
6. The subject does not have a known allergy to chicken eggs or a history of a severe reaction to an influenza vaccination in the past.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2005-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
- Rate of influenza immunization among subjects

SECONDARY OUTCOMES:
Change in knowledge, attitutes, and beliefs regarding influenza and influenza immunization.
Changes in health behaviors around influenza (e.g. hand washing and cough etiquette).
General health outcomes related to respiratory illnesses (e.g. number of influenza-like illnesses, number of physician visits, number of missed work days).
Rate of influenza immunization among subject household members.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Mandl, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nichol KL. Cost-benefit analysis of a strategy to vaccinate healthy working adults against influenza. Arch Intern Med. 2001 Mar 12;161(5):749-59. doi: 10.1001/archinte.161.5.749. PMID 11231710
- [Background] Keech M, Scott AJ, Ryan PJ. The impact of influenza and influenza-like illness on productivity and healthcare resource utilization in a working population. Occup Med (Lond). 1998 Feb;48(2):85-90. doi: 10.1093/occmed/48.2.85. PMID 9614766
- [Background] Harper SA, Fukuda K, Uyeki TM, Cox NJ, Bridges CB; Advisory Committee on Immunization Practices (ACIP), Centers for Disease Control and Prevention (CDC). Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2005 Jul 29;54(RR-8):1-40. PMID 16086456
- [Background] Bridges CB, Thompson WW, Meltzer MI, Reeve GR, Talamonti WJ, Cox NJ, Lilac HA, Hall H, Klimov A, Fukuda K. Effectiveness and cost-benefit of influenza vaccination of healthy working adults: A randomized controlled trial. JAMA. 2000 Oct 4;284(13):1655-63. doi: 10.1001/jama.284.13.1655. PMID 11015795
- [Background] Mandl KD, Szolovits P, Kohane IS. Public standards and patients' control: how to keep electronic medical records accessible but private. BMJ. 2001 Feb 3;322(7281):283-7. doi: 10.1136/bmj.322.7281.283. No abstract available. PMID 11157533
- [Background] Riva A, Mandl KD, Oh DH, Nigrin DJ, Butte A, Szolovits P, Kohane IS. The personal internetworked notary and guardian. Int J Med Inform. 2001 Jun;62(1):27-40. doi: 10.1016/s1386-5056(00)00136-2. PMID 11340004
- [Background] Mandl KD, Overhage JM, Wagner MM, Lober WB, Sebastiani P, Mostashari F, Pavlin JA, Gesteland PH, Treadwell T, Koski E, Hutwagner L, Buckeridge DL, Aller RD, Grannis S. Implementing syndromic surveillance: a practical guide informed by the early experience. J Am Med Inform Assoc. 2004 Mar-Apr;11(2):141-50. doi: 10.1197/jamia.M1356. Epub 2003 Nov 21. PMID 14633933
- [Background] Heffernan R, Mostashari F, Das D, Karpati A, Kulldorff M, Weiss D. Syndromic surveillance in public health practice, New York City. Emerg Infect Dis. 2004 May;10(5):858-64. doi: 10.3201/eid1005.030646. PMID 15200820
- [Derived] Bourgeois FT, Simons WW, Olson K, Brownstein JS, Mandl KD. Evaluation of influenza prevention in the workplace using a personally controlled health record: randomized controlled trial. J Med Internet Res. 2008 Mar 14;10(1):e5. doi: 10.2196/jmir.984. PMID 18343794